CLINICAL TRIAL: NCT01546948
Title: Intraoperative Opioids and Postoperative Recovery After Hepatobiliary or Foregut Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH11-232
Record Dates: First submitted 2012-03-03; First posted 2012-03-07 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Pain
Keywords: Methadone; Hydromorphone; Hepatobiliary surgery; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Patients in the methadone group will be administered 0.3 mg/kg of methadone intraoperatively: two-thirds of the dose (6 cc or 0.2 mg/kg of methadone) on induction of anesthesia as a bolus. The remainder of the dose (3 cc or 0.1 mg/kg of methadone) will be administered at approximately 1.5-2 hours before the end of the procedure.
  Interventions: Drug: Methadone
- Hydromorphone (Active Comparator): Patients in the hydromorphone group will receive 0.03 mg/kg of hydromorphone; two-thirds the dose (6 cc or 0.02 mg/kg) on induction of anesthesia, and the remainder of the hydromorphone (3 cc or 0.01 mg/kg) will be bolused 1.5-2 hours before surgery concludes.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Methadone — Patients in the methadone group will be administered 0.3 mg/kg of methadone intraoperatively: two-thirds of the dose (6 cc or 0.2 mg/kg of methadone) on induction of anesthesia as a bolus. The remainder of the dose (3 cc or 0.1 mg/kg of methadone) will be administered at approximately 1.5-2 hours before the end of the procedure.
  Arms: Methadone
Drug: Hydromorphone — Patients in the hydromorphone group will receive 0.03 mg/kg of hydromorphone; two-thirds the dose (6 cc or 0.02 mg/kg) on induction of anesthesia, and the remainder of the hydromorphone (3 cc or 0.01 mg/kg) will be bolused 1.5-2 hours before surgery concludes.
  Arms: Hydromorphone

SUMMARY:
The primary aim of this randomized, double-blind study is to examine the effect of a single intraoperative dose of methadone on analgesic requirements during the first three days after hepatobiliary or foregut surgery. These patients will be compared to subjects receiving a standard dose of the "traditional" intraoperative opioid (hydromorphone). Secondary outcome measures to be assessed will include postoperative pain scores and standard recovery variables such as hospital length of stay.

DETAILED DESCRIPTION:
60 patients will be enrolled in this clinical trial. All patients presenting for elective hepatobiliary or foregut surgery will be eligible for enrollment.

Patients will be randomized to receive either methadone or hydromorphone on the basis of a computer generated random number table. Patients in each group will receive standard clinical intraoperative doses of either methadone (0.3 mg/kg) or hydromorphone (0.03 mg kg). These doses (0.3 mg/kg of methadone or 0.03 mg/kg of hydromorphone) represent dosages which appear to be approximately equipotent. Study medications will be prepared by the pharmacy in 10 cc syringes, and all clinicians will be blinded to group assignment Patients in the methadone group will be administered two-thirds of the dose (6 cc or 0.2 mg/kg of methadone) on induction of anesthesia as a bolus. The remainder of the dose (3 cc or 0.1 mg/kg of methadone) will be administered at approximately 1.5-2 hours before the end of the procedure. In the hydromorphone group, patients will receive two-thirds the dose (6 cc or 0.02 mg/kg) on induction of anesthesia, and the remainder of the hydromorphone (3 cc or 0.01 mg/kg) will be bolused 1.5-2 hours before surgery concludes. All other anesthestic management will be standardized.

Data Collection The primary endpoint of the study is total dose of intravenous hydromorphone used during the first 3 days after surgery. A blinded research assistant will record the total doses of hydromorphone used in the PACU and with the PCA device during the first 24, 48, and 72 hour after surgery. Several secondary endpoints will be evaluated. Pain in the postoperative period will be assessed at several time points; PACU arrival, 1, 2, 4, and 8 hours after surgery, and then approximately 8 AM and 4 PM on postoperative days 1-3. Pain will be quantified by a blinded research assistant using an 11-point verbal rating scale (0=no pain, 10=worst pain imaginable). Pain will be determined at rest and with coughing. The presence or absence of nausea and vomiting will be determined. Level of sedation will be measured by observers using a 4-point sedation scale (0=fully awake, 1=mildly sedated (seldom drowsy and easy to awake, 2=moderately sedated (often drowsy and easy to awake), 3=severely sedated (somnolent, difficult to awake).

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective hepatobiliary or foregut surgery will be eligible for enrollment

Exclusion Criteria:

* Exclusion criteria include:

  1. Preoperative renal failure (defined as a serum creatinine > 2.0 mg/dL.)
  2. Morbid obesity
  3. American Society of Anesthesiologists Physical Status IV or V
  4. Age > 80 years
  5. Pulmonary disease necessitating home oxygen therapy
  6. Allergy to methadone or hydromorphone
  7. Preoperative recent history of opioid or alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain medication used (hydromorphone) | First 72 hours after surgery
  A blinded research assistant will record the total doses of hydromorphone used in the PACU and with the PCA device during the first 24, 48, and 72 hour after surgery.

SECONDARY OUTCOMES:
Postoperative pain scores | First 72 hours after sugery
  Pain in the postoperative period will be assessed at several time points; PACU arrival, 1, 2, 4, and 8 hours after surgery, and then approximately 8 AM and 4 PM on postoperative days 1-3. Pain will be quantified by a blinded research assistant using an 11-point verbal rating scale (0=no pain, 10=worst pain imaginable). Pain will be determined at rest and with coughing.
The presence or absence of nausea and vomiting | First 72 hours after surgery
  The presence or absence of nausea and vomiting will be determined by a blinded research assistant
Level of sedation | First 72 hours after surgery
  Level of sedation will be measured by observers using a 4-point sedation scale (0=fully awake, 1=mildly sedated (seldom drowsy and easy to awake, 2=moderately sedated (often drowsy and easy to awake), 3=severely sedated (somnolent, difficult to awake).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States